## **Study Identification**

ClinicalTrials.gov ID: NCT03119025

Brief Title: Autologous Dendritic Cell Vaccine for Treatment of Patients with Chronic

**HCV-Infection** 

Name of Researcher

Signature

April 10, 2015

## Informed Consent Form for Research Involving Human Subjects

You are being invited to participate in a research study, which the Institute of Fundamental and Clinical Immunology (IFCI) Institutional Review Board (IRB) has reviewed and approved (approval no 88, 04/10/2015). This form is designed to provide you - as a human subject - with information about this study. The Investigator will describe this study to you and answer any of your questions. You are entitled to a copy of this form. If you have any questions or complaints about the informed consent process of this research study or your rights as a subject, please contact the IRB at the IFCI Office of Institutional Research at (383) 228-54-21 or <a href="mailto:cke@nqs.ru">cke@nqs.ru</a>.

Thank you for agreeing to participate in this research project.

**Project Title:** Safety/Efficacy of Vaccination With Autologous Dendritic Cells Pulsed With Recombinant HCV-Antigens (Core and NS3) for Treatment of Patients With Chronic HCV-Infection

Principal Investigator: Alexander A Ostanin, PhD, MD, Head of Clinical Department, (383) 236-03-29

I, the undersigned, confirm that (please tick box as appropriate):

| 1. | I have read and understood the information about the project, as provided in the Information<br>Sheet |
|---|---|
| 2. | I have been given the opportunity to ask questions about the project and my participation. |
| 3. | I voluntarily agree to participate in the project. |
| 4. | I understand I can withdraw at any time without giving reasons and that I will not be penalized for withdrawing nor will I be questioned on why I have withdrawn. |
| 5. | The procedures regarding confidentiality have been clearly explained (e.g. use of names, pseudonyms, anonymisation of data, etc.) to me. |
| 6. | If applicable, separate terms of consent for interviews, audio, video or other forms of data collection have been explained and provided to me. |
| 7. | The use of the data in research, publications, sharing and archiving has been explained to me. |
| 8. | I understand that other researchers will have access to this data only if they agree to preserve the confidentiality of the data and if they agree to the terms I have specified in this form. |
| 9. | Select only <b>one</b> of the following: I would like my name used and understand what I have said or written as part of this study will be used in reports, publications and other research outputs so that anything |
| | I have contributed to this project can be recognised. I do not want my name used in this project. |
| 10. | I, along with the Researcher, agree to sign and date this informed consent form. |
| Participant: Name of Participant Signature Date Researcher: | |

Date